CLINICAL TRIAL: NCT05326204
Title: 1 Versus 2 Hours Post Meal Self Monitoring Blood Glucose in Gestational Diabetes Mellitus on Treatment-A Prospective Randomised Controlled Trial
Brief Title: 1 Versus 2 Hours Post Meal Glucose Monitoring in Gestational Diabetes on Treatment
Status: Recruiting | Type: Observational
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Other Study IDs: FF-2022-002
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Gestational Diabetes; Treatment Adherence
Keywords: Gestational diabetes; treatment; glucose monitoring
MeSH Terms: conditions — Diabetes, Gestational; Treatment Adherence and Compliance | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1 hour: Blood glucose monitoring comprises of 1 hour post meal
  Interventions: Other: Home blood glucose monitoring
- 2 hours: Blood glucose monitoring comprises of 2 hours post meal
  Interventions: Other: Home blood glucose monitoring

INTERVENTIONS:
Other: Home blood glucose monitoring — Self monitoring of capillary blood glucose

SUMMARY:
A study to compare between 1 and 2 hours post meal blood glucose monitoring in patients with Gestational Diabetes Mellitus requiring treatment.

DETAILED DESCRIPTION:
This study involves all pregnant women who attended our antenatal clinic with Gestational Diabetes Mellitus requiring treatment. They will be randomised to either 1 or 2 hours post meal self blood glucose monitoring. The blood sugar profile is a staggered 7 points. They are followed up in the research clinic until delivery.

ELIGIBILITY:
Inclusion Criteria:

* Gestational diabetes diagnosed based on National Institute for Health and Care Excellence guideline
* requiring treatment either with metformin alone or combined with insulin

Exclusion Criteria:

* type 1 and 2 diabetes
* bad obstetrics history
* underlying medical disorders such as Systemic Lupus Erythematosus
* fetal anomaly
* delivery elsewhere

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All women with gestational diabetes on treatment attending the antenatal clinic in our centre
Sampling Method: Non-Probability Sample
Enrollment: 2954 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2025-12-29 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Mode of delivery | from point of randomization to birth of the neonate
  route
Gestational age | from point of randomization to birth of the neonate
  in weeks
Fetal weight | from point of randomization to birth of the neonate
  in gram

SECONDARY OUTCOMES:
Maternal complications | from point of randomization to birth of the neonate
  postpartum haemorrhage, perineal tear
perinatal complications | from point of randomization to birth of the neonate
  intrauterine death, macrosomia, admission to neonatal intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Rahana Abd Rahman, Principal Investigator — National University of Malaysia
Locations (1):
- UKM Medical Center, Kuala Lumpur, W.Persekutuan, Malaysia

IPD SHARING:
Plan to Share IPD: No